CLINICAL TRIAL: NCT00935714
Title: Exercise and Breast Cancer Related Lymphedema: Influence of Muscle Group and Sequence on Volume Change in Swollen and Normal Arms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Prof. A. Sternberg, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 0023-09-HYMC
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Arm; Lymphedema; Breast Cancer; Exercise; Breast Cancer related Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Motor Activity; Breast Cancer Lymphedema | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Muscle Group (Active Comparator): Exercise
  Interventions: Other: Exercise
- Sequence (Active Comparator): Exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise
  Arms: Muscle Group
Other: Exercise
  Arms: Sequence

SUMMARY:
Arm exercise influences arm volume and symptoms in breast cancer related lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* unilateral arm lymphedema as a result of breast cancer treatment
* completion of breast cancer treatments
* arm lymphedema onset 3 months or more after surgery and persistent for at least 6 months
* in the maintenance phase of lymphedema treatment

Exclusion Criteria:

* women with recurrent cancer
* intercurrent diseases affecting the swollen arm
* lack of understanding of the Hebrew language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Improved arm volume measurement | Weekly for five weeks

SECONDARY OUTCOMES:
Quality of Life | Weekly for 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel